CLINICAL TRIAL: NCT02400294
Title: Prevention of Ventilator Associated Pneumonia With Toothbrushing in Oral Care of Critically Ill Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0227
Record Dates: First submitted 2015-03-16; First posted 2015-03-27 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Critical Care; Mechanical Ventilation; Ventilator Associated Pneumonia Prevention; Toothbrushing; Oral Care
Keywords: Critical care; Mechanical ventilation; Ventilator associated pneumonia; Oral care
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Toothbrushing

STUDY DESIGN:
Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: Toothbrushing — Toothbrushing associated with standard oral care in mechanically ventilated patients

SUMMARY:
Effect of toothbrushing in oral care of mechanically ventilated critically ill patients on prevention of ventilator associated pneumonia

DETAILED DESCRIPTION:
Prospective, before and after study in 5 Intensive Care Units (ICUs) of a university hospital.

The before period (control phase, 6 months): standard oral care 3 times a day in every consecutive intubated patients in the participating ICUs The interphase period (1 month): formal training of all the nurses, physicians and residents on the use of toothbrushing during oral care The after period: (study phase, 6 months): standard oral care with tooth brushing 3 times a day in every consecutive intubated patients in the participating ICUs

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Intubated mechanically ventilated ICU patient
* Platelets count >50G/L

Exclusion Criteria:

* Edentulous patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 2030 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Nosocomial ventilator associated pneumonia | at Day-28
  Presence of at least two signs (body fever greater than 38°C; leukocytosis greater than 12000/ml or leukopenia below 4000/ml, purulent pulmonary secretions) associated with the appearance of a new infiltrate or modification of an existing infiltrate on chest-X-ray. Confirmation by a lower respiratory tract sample using a quantitative culture with a predefined positive threshold. Hospital-acquired pneumonia was defined as a pneumonia that occurs at least 48 hours after admission, which was not incubating at time of admission (Am J Respir Crit Care Med 2005; 171, 388-416).

SECONDARY OUTCOMES:
Tracheobronchitis | at Day-28
  Association of at least two signs (fever above 38.0°C, Leucocytosis above 12000/ml or purulent pulmonary secretions) with isolation of bacteria in a lower respiratory tract sample without modification of chest-X-Ray.
ICU length of stay | at Day-90
ICU mortality | at Day-90
Hospital mortality | at Day-90
Antibiotic free days | at Day-90

CONTACTS AND LOCATIONS:
Overall Officials: Russel CHABANNE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Ory J, Mourgues C, Raybaud E, Chabanne R, Jourdy JC, Belard F, Guerin R, Cosserant B, Faure JS, Calvet L, Pereira B, Guelon D, Traore O, Gerbaud L. Cost assessment of a new oral care program in the intensive care unit to prevent ventilator-associated pneumonia. Clin Oral Investig. 2018 Jun;22(5):1945-1951. doi: 10.1007/s00784-017-2289-6. Epub 2017 Nov 30. PMID 29189950